CLINICAL TRIAL: NCT02562092
Title: The Georgia Latino AIDS/HIV Diagnosis and Linkage in Youth (GLADLY) Project
Acronym: GLADLY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was not able to be completed due to the COVID-19 pandemic.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Andres Camacho-Gonzalez, Assistant Professor of Pediatrics, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00080817
Record Dates: First submitted 2015-09-24; First posted 2015-09-29 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: HIV
Keywords: AIDS; Health Promotion
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Palliative Care; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Focus Group (No Intervention): Participants will complete a questionnaire and will be involved in a group discussion regarding good sites within the community to perform HIV testing.
- Venue Testing Group- Negative Test (Other): Participants will perform a rapid HIV test and will be asked to answer questions about their sexual life and living situation. No followup is needed for a negative HIV test.
  Interventions: Behavioral: Reducing Risk Behavior
- Venue Testing Group- Positive Test (Other): Participants will perform a rapid HIV test and will be asked to answer questions about their sexual life and living situation. Participants with a positive HIV test will receive care from a psychologist and case manager for one year.
  Interventions: Behavioral: Support and Guidance

INTERVENTIONS:
Behavioral: Reducing Risk Behavior — A small survey will be conducted to identify risk factors and assess demographics. Participants will receive psychological support and counseling on reducing risk behavior for one year.
  Arms: Venue Testing Group- Negative Test
Behavioral: Support and Guidance — A small survey will be conducted to identify risk factors and assess demographics. Participants with a positive HIV test will receive standard HIV care, support, and guidance from a psychologist and case manager including an assessment of basic needs (food, clothing, shelter), and counseling on risk taking behaviors for one year.
  Arms: Venue Testing Group- Positive Test

SUMMARY:
This study aims to understand the barriers to receiving HIV testing and retention of care for at risk and HIV positive young adults. This study also seeks to determine the feasibility and acceptability of HIV testing in a non-clinical setting.

DETAILED DESCRIPTION:
This study aims to identify factors that can facilitate or impede the use of non-clinical HIV testing venues as well as identify potential testing sites and assess acceptability of an HIV prevention intervention. In addition, the study will implement a pilot intervention to test the feasibility non-clinical HIV testing and follow up events for HIV positive youth.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active
* HIV positive or negative
* Latino youth ages 18-24 years
* Residents of the state of Georgia and can understand spoken and written English or Spanish.

Exclusion Criteria:

* Unmet inclusion criteria

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2015-08; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Days to Linkage to Care | Post Diagnosis (Up to 3 months)
  For participants who test positive, linkage to care is measured as the number of days to seek HIV treatment.

SECONDARY OUTCOMES:
Number of medical care visits | Post Diagnosis (Up to one year)
  For participants who test positive, engagement to care is measured as the number of medical care visits in a six month period after diagnosis. One HIV medical care visit every six months is considered engaged.
Change in CD4 count | Baseline (Post Diagnosis), One year assessment (Up to one year)
  A CD4 count is a lab test that measures the number of CD4 T lymphocytes (CD4 cells) in a blood sample. A very low CD4 count (less than 200 cells/mm3) is a way to determine whether an HIV infection has progressed. Change is measured as the difference in CD4 count from baseline to the end of the study period.
Change in viral load | Baseline (Post Diagnosis), One year assessment (Up to one year)
  A viral load test is a lab test that measures the number of HIV virus particles in a milliliter of blood. A high viral load indicates the presence of more HIV within the body. Change is measured as the difference in viral load from baseline to the end of the study period.
Rate of venue acceptance | One year assessment (Up to one year)
  The rate of venue acceptance is measured as the number of venues that allow rapid HIV testing over he number of venues approached.
Rate of study subject acceptance | One year assessment (Up to one year)
  The rate of study subject acceptance is measured as the number of participants who agree to participate in rapid HIV testing over the number of people approached.
Change in HIV stigma scale score | Baseline (Post Diagnosis), One year assessment (Up to one year)
  The HIV stigma scale is a ten question self report measure that assesses perceived feelings of being stigmatized. Answers are reported on a scale from 0 (not at all) to 4 (extremely). A higher score indicates feelings of greater stigmatization.
Change in HIV-AIDS stress scale score | Baseline (Post Diagnosis), One year assessment (Up to one year)
  The HIV-AIDS stress scale is a self report measure that assesses perceived emotional stress related to HIV. Answers are reported on a scale from 0 (not at all) to 4 (extremely). A higher score indicates more emotional stress.

CONTACTS AND LOCATIONS:
Overall Officials: Andres Camacho-Gonzalez, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Health System, Atlanta, Georgia
  - Ponce De Leon Center, Atlanta, Georgia